CLINICAL TRIAL: NCT05345938
Title: A Phase I/II Study to Evaluate the Safety, Tolerability, Efficacy, and Pharmacokinetics of Mitoxantrone Hydrochloride Liposome Injection in Subjects With Acute Myeloid Leukemia
Brief Title: A Study of Mitoxantrone Hydrochloride Liposome Injection in Subjects With Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Adjust the research strategy.
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HE071-029
Record Dates: First submitted 2022-04-06; First posted 2022-04-26 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2022-01

CONDITIONS: Relapsed or Refractory Acute Myeloid Leukemia (AML)
MeSH Terms: conditions — Recurrence; Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mitoxantrone Hydrochloride Liposome Injection (Experimental): Stage 1: Subjects with R/R AML will receive one of three dose-escalation (30 mg/m^2, 36 mg/m^2, 40 mg/m^2) Mitoxantrone Hydrochloride Liposome, IV, on day 1 of each 28-day cycle (q4w).
  Stage 2: Subjects with R/R AML or unfit AML will receive one dose Mitoxantrone Hydrochloride Liposome every 28 days (a cycle) for a maximum of 6 cycles.
  Interventions: Drug: Mitoxantrone Hydrochloride Liposome

INTERVENTIONS:
Drug: Mitoxantrone Hydrochloride Liposome — Intravenous injection (IV), on day 1 of each 28-day cycle (q4w)
  Other Names: HE071

SUMMARY:
This is a multi-center, open-label, single-arm, phase I/II study to evaluate the safety, tolerability, efficacy, and pharmacokinetics of mitoxantrone hydrochloride liposome injection in subjects with acute myeloid leukemia (AML).

DETAILED DESCRIPTION:
This study will have two stages. Stage 1: Dose escalation, about 9-18 subjects, who are either refractory to induction therapy or have relapsed (R/R) after achieving remission with prior therapy will be recruited. The enrolled subjects will receive Mitoxantrone Hydrochloride Liposome injection in one of three dose-escalation (30 mg/m^2, 36 mg/m^2, 40 mg/m^2) by intravenous infusion (IV), every 28 days (q4w, 1 cycle). If the patient achieves remission (at least PR) after at most 2 cycles of induction, the original regimen of consolidation therapy can be continued for 2-4 cycles, with a total course of no more than 6 cycles. The DLT observation period is 28 days after the first dose in cycle 1, and including the first 28 days treatment cycle. Subjects in Cycle 1 will have PK sampling performed. Stage 2: Dose expansion, about 35-72 subjects with R/R AML or unfit AML will be recruited. The subjects will receive Mitoxantrone Hydrochloride Liposome dose according to the results of stage 1. If the patient achieves remission (at least PR) after at most 2 cycles of induction, the original regimen of consolidation therapy can be continued for 2-4 cycles, with a total course of no more than 6 cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects fully understand, voluntarily participate in this study and sign the informed consent form;
2. Age ≥18 years old, male or female;
3. Morphological and/or pathological confirmation of relapsed/refractory AML after prior anti-leukemic therapy or newly diagnosed unfit AML (dose expansion stage) , which are judged by the investigator to be unsuitable for intensive chemotherapy;
4. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 2 for subjects with R/R AML or aged over 75 years old, 0-3 for subjects with unfit AML aged 18 to 74 years old;
5. The organ function level must meet the following requirements:

Liver function : Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3 times normal upper limit (ULN); Total bilirubin ≤1.5 x ULN ( ≤ 3.0 x ULN for subjects with unfit AML); Renal function: Blood creatinine ≤1.5 x ULN (creatinine clearance <45 mL/min for subjects with unfit AML); 6. Subjects and their partners agree to take effective contraception from the date of signing an informed consent to 6 months after the last dose (for example: combined hormone (contain estrogen and progesterone), combining inhibit ovulation, progestin contraception and inhibit ovulation, intrauterine device, intrauterine hormone release system, bilateral vasectomy, bilateral tubal ligation, avoiding sexual behavior, etc.); female subjects must have negative blood HCG (except menopause, hysterectomy or bilateral oophorectomy).

Exclusion Criteria:

1. AML occurs in any of the following situations:

1. Acute promyelocytic leukemia;
2. Chronic myeloid leukaemia in blast crisis;
3. Central nervous system (CNS) involvement with AML; 2. Subjects has been previously diagnosed with other malignant tumors in the past 5 years (except curable tumors such as basal cell carcinoma of the skin and carcinoma in situ of the cervix); 3. Graft-versus-host disease requiring ongoing treatment and having received more than one allogeneic stem cell transplant.

4. History of allergy to mitoxantrone hydrochloride injection or liposomal drugs; 5. Previous treatment with doxorubicin or other anthracycline and a cumulative dose of doxorubicin in excess of 400mg/m^2 (anthracycline equivalent dose calculation: 1 mg doxorubicin =2 mg epirubicin = 2 mg daunorubicin = 0.5 mg idarubicin = 0.45 mg mitoxantrone; Adriamycin liposomes excepted); 6. Received any antineoplastic therapy within 2 weeks prior to initial administration (or within 5 half-lives of the drug). Except for leukocyte lowering therapy (hydroxyurea, leukocyte separation, etc.) and prophylactic intrathecal injection which are over 24 hours prior to administration; 7.The non-hematologic toxicity of previous anti-tumor treatment > Grade 1 based on CTCAE (except for alopecia, skin pigmentation or tolerable events judged by the investigator); 8. Those on systemic anti-infective therapy with poorly controlled infection (signs of infection progression within 1 week prior to the first dose, or as determined by the investigator); 9. Life expectancy < 3 months; 10. Cardiovascular diseases, including but not limited to:

1. QTc interval >480 ms or long QTc syndrome in screening;
2. Complete left bundle branch block, severe atrioventricular block (without pacemaker);
3. Requiring treatment of serious and uncontrolled arrhythmias, unstable angina pectoris, valvular disease, etc;
4. Have a history of chronic congestive heart failure, New York Heart Association（NYHA）≥3; or persistent cardiomyopathy;
5. Uncontrolled hypertension (defined as multiple measurements of systolic blood pressure >150 mmHg or diastolic blood pressure >90 mmHg under medication control);
6. ECG evidence of myocardial infarction, viral myocarditis, history of severe pericardial disease, acute ischemic or active conduction system abnormalities within 6 months prior to screening; 11. Severe thrombosis or thromboembolism in the past 6 months, including but not limited to cerebrovascular accident (including transient ischemic attack, etc.), upper/lower vena cava thrombosis, lower extremity deep vein thrombosis, pulmonary embolism, etc; 12. HBsAg or HBcAb positive, with HBV DNA≥2000 IU/mL, or HCV antibody positive with HCV RNA higher than the lower limit of the detection value of the research center, or HIV antibody positive in the preliminary screening; 13. Subjects are suffering from any other serious and/or uncontrollable disease that, in the judgment of the investigator, may affect the patient's participation in this study (including but not limited to: uncontrolled diabetes, kidney disease requiring dialysis treatment, severe liver diseases, life-threatening autoimmune disease and hemorrhagic disease, drug abuse, nervous system diseases, etc.); 14. Pregnant or lactating female; 15. Not suitable for this study as decided by the investigator due to other reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-06-14 (Actual); Primary Completion 2022-11-19 (Actual); Study Completion 2022-11-19 (Actual)

PRIMARY OUTCOMES:
DLT | At the end of Cycle 1 (each cycle is 28 days)
  Number of Participants with Dose Limiting Toxicities (DLTs, Stage 1)
CR | From the initiation of the first dose to 28 days after the last dose
  Complete remission (CR) rate (Stage 2)

SECONDARY OUTCOMES:
TEAEs | From the initiation of the first dose to 28 days after the last dose
  Treatment-emergent adverse events (TEAEs)
CR rate | From the initiation of the first dose to 28 days after the last dose
  CR rate (Stage 1)
CRc | At the end of Cycle 2 (each cycle is 28 days)
  Composite complete response (CRc) rate CRc includes CR and CR with incomplete blood recovery (CRi).
ORR | At the end of Cycle 2 (each cycle is 28 days)
  Objective response rate (ORR) Objective response includes CR, CR with CRi , morphologic leukemia-free status (MLFS) and partial remission (PR).
EFS | up to 36 months
  Event--free survival (EFS)
OS | From the enrollment to the death of last subject or the end of the clinical trial (up to 36 months)
  Overall survival (OS)
Tmax | Within 1hour before IV administration of the first cycle to 1hour before the second cycle
  Peak time (Tmax)
Cmax | Within 1hour before IV administration of the first cycle to 1hour before the second cycle
  Maximum concentration (Cmax) of Mitoxantrone Hydrochloride Liposome
AUC0-t | Within 1hour before IV administration of the first cycle to 1hour before the second cycle
  Area Under the Concentration-Time Curve from Time Zero to Last Measurable Concentration (AUC0-t) of Mitoxantrone Hydrochloride Liposome
AUC0-∞ | Within 1hour before IV administration of the first cycle to 1hour before the second cycle
  Area Under the Concentration-Time Curve from Time Zero to Last Measurable Concentration (AUC0-∞) of Mitoxantrone Hydrochloride Liposome
t1/2 | Within 1hour before IV administration of the first cycle to 1hour before the second cycle
  Half-time (t1/2） of Mitoxantrone Hydrochloride Liposome
CL | Within 1hour before IV administration of the first cycle to 1hour before the second cycle
  Clearance ( CL) of Mitoxantrone Hydrochloride Liposome
Vz | Within 1hour before IV administration of the first cycle to 1hour before the second cycle
  Apparent Volume of Distribution ( Vz) of Mitoxantrone Hydrochloride Liposome

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China